CLINICAL TRIAL: NCT00798668
Title: The Body's Response to Food Intake in Trained, Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Wayne Campbell, Professor, Foods and Nutrition, Purdue University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0607004184; NIH R01 AG021911-0102
Record Dates: First submitted 2008-11-25; First posted 2008-11-26 (Estimated); Last update posted 2013-09-24 (Estimated); Status verified 2010-03

CONDITIONS: Elderly
Keywords: Endocrine and Gastrointestinal Response to Food

ARMS (4):
- 1 (Experimental): participants continue current exercise and take liquid supplement
  Interventions: Dietary Supplement: Liquid Supplements
- 2 (Experimental): Participants continue current exercise and take solid supplement
  Interventions: Dietary Supplement: Solid Supplement
- 3 (Experimental): Participants continue current sedentary behavior and take liquid supplements
  Interventions: Dietary Supplement: Liquid Supplements
- 4 (Experimental): Participants continue current sedentary behavior and take solid supplements
  Interventions: Dietary Supplement: Solid Supplement

INTERVENTIONS:
Dietary Supplement: Liquid Supplements — Liquid supplement that provides 12.5% of the subjects total energy requirement.
  Arms: 1; 3
Dietary Supplement: Solid Supplement — Solid supplement that provides 12.5% of the subjects total energy requirement.
  Arms: 2; 4

SUMMARY:
The purpose of this research study is to determine the effects of food supplements and strength training on appetite, the amount of energy expended, and body composition.

ELIGIBILITY:
Inclusion Criteria:

All subjects must meet the following eligibility criteria:

* Age range: 60 years and older
* Body mass index between 20-29 kg/m2
* Weight stable (< 2 kg weight change within last 6 months)
* Non-smoking
* Constant habitual activity patterns within last 3 months
* Clinically normal blood profiles (specifically, normal liver and kidney function; normal complete blood count (non-anemic); fasting blood glucose <110 mg/dl)
* Not taking medications known to influence appetite or metabolism
* Non-diabetic
* Confirmation of acceptability of eating the study test foods (solids and fluids)

Trained subjects (Recruiting 36; N-25) must meet the following eligibility criteria:

* Resistive exercise training (≥ 2 times a week) based on reported physical activity levels (questionnaire)
* Active fitness level (≥ 2, 30-minute aerobic exercise sessions/week)

Sedentary subjects (Recruiting 36; N-25) must meet the following eligibility criteria:

* Resistive exercise training (≤ 1 time a week) based on reported physical activity levels (questionnaire)
* Active fitness level (≤ 2, 30-minute aerobic exercise sessions/week)

Exclusion Criteria:

All subjects will be excluded based on the following exclusionary criteria:

* Age: <60 years
* Body mass index: outside of the 20-29 kg/m2 range
* Gained or lost > 4.5 kg within the last 6 months
* Smoker (currently or within the last year)
* Intermittently been involved in a diet and/or exercise program within the last 3 months
* Clinically abnormal blood profiles as identified by our study physician, Arthur Rosen, MD
* Taking medications (currently or within the last 3 months) known to influence appetite or metabolism
* Abnormal heart function (interpreted by a cardiologist) and assessed (for study exclusion) by our study physician, Arthur Rosen, MD
* Clinically diagnosed as diabetic
* Study foods are found to be unacceptable for consumption by the subject
* Clinically diagnosed osteoporosis

Trained subjects will be excluded based on the following exclusionary criteria:

* Did not perform resistive exercise training (currently or within the last 3 months) based on reported physical activity levels (questionnaire)
* Perform ≤ 1, 30-minute aerobic exercise session/week (currently or within the last 3 months) based on physical activity levels questionnaire)

Sedentary subjects will be excluded based on the following exclusionary criteria:

* Performed resistive exercise training (currently or within the last 3 months) based on reported physical activity levels (questionnaire)
* Perform > 2, 30-minute aerobic exercise sessions/week (currently or within the last 3 months) based on physical activity levels questionnaire)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-09; Primary Completion 2007-08 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Quantify the acute effects of fluid and solid foods on post-prandial (post-meal) appetite and food intake at the next eating occasion in trained and untrained, elderly people. | 6 weeks

SECONDARY OUTCOMES:
Quantify the contribution of selected satiety factors (glucose, insulin, CCK, ghrelin, and GLP-1) and gastrointestinal transit time, to the differential appetitive responses to fluid versus solid foods in trained and untrained, elderly people | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Purdue University, West Lafayette, Indiana, United States